CLINICAL TRIAL: NCT01563081
Title: A Multi-Center, Open-labelled Study to Evaluate the Safety of Levocetirizine Hydrochloride Oral Solution in Children Aged 6 Months to 2 Years With Allergic Rhinitis or Pruritus Associated With the Skin Diseases.
Brief Title: Safety Study of Levocetirizine Oral Solution for Japanese Pediatrics
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 116455
Record Dates: First submitted 2012-03-15; First posted 2012-03-26 (Estimated); Results first posted 2013-06-03 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2017-01

CONDITIONS: Rhinitis
Keywords: Allergic rhinitis; Pediatric; Pruritus; Levocetirizine
MeSH Terms: conditions — Rhinitis; Rhinitis, Allergic; Pruritus | interventions — levocetirizine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Levocetirizine (Experimental): Clear solution, 0.50 mg levocetirizine dihydrochloride contains in one milliliter of the solution
  Interventions: Drug: Levocetirizine

INTERVENTIONS:
Drug: Levocetirizine — Clear solution, 0.50 mg levocetirizine dihydrochloride contains in one milliliter of the solution. Levocetirizine oral solution are administered once daily at a dose of 2.5 mL (1.25 mg of levocetirizine) in the morning to infants aged between 6 months and 1 year old
Drug: Levocetirizine — Clear solution, 0.50 mg levocetirizine dihydrochloride contains in one milliliter of the solution. Levocetirizine oral solution are administered twice daily at a dose of 2.5 mL (1.25 mg of levocetirizine) in the morning and evening before sleep to infants aged between 1 year and 2 years old

SUMMARY:
To evaluate the safety of treatment with levocetirizine oral solution in pediatric patients aged form 6 months to 2 years old with allergic rhinitis or pruritus associated with the skin diseases.

DETAILED DESCRIPTION:
This is a multi-center, open-labelled study to confirm the safety as main objective, and consisting of minimum 1-week screening period and 2-week treatment period. The subjects who meet the inclusion criteria are to be placed on one of the following two regimens according to their ages at the start of treatment period: once daily administration of levocetirizine at a dose of 1.25 mg (in the morning) to infants aged between 6 months and 1 year old (younger age group), and twice daily administration of levocetirizine at a dose of 1.25 mg (in the morning, in the evening before sleep) to infants aged between 1 year and 2 years old (older age group).

ELIGIBILITY:
Inclusion Criteria:

* Outpatients
* Either boys or girls are acceptable.
* Pediatric patients ranging from 6 months to 2 years in age at the time of initiation of the treatment in clinical trial
* Pediatric patients who have at least one of the symptoms associated with allergic rhinitis including rhinorrhea, nasal congestion and sneezing, and require at least 2-week treatment with antihistamine drugs, or those who suffer from pruritus associated with the following diseases and require at least 2-week treatment with antihistamine drugs (- Chronic urticaria, - Eczema/dermatitis group: atopic dermatitis etc. [A diagnosis of atopic dermatitis is made in accordance with the "Definition/Diagnostic Criteria of Atopic Dermatitis, - Prurigo group: acute prurigo (strophulus, urticaria-like lichen, etc.), subacute prurigo, chronic prurigo (nodular prurigo etc.), - Pruritus cutaneous: systemic pruritus cutaneous, local pruritus cutaneous)
* Pediatric patients with QTc interval below 450 msec. QTc interval shall be below 480 msec in the pediatric patients with bundle branch block at screening (A judgment shall be made according to the QTc interval based on ECG result corresponding to one heart beat or the QTc interval based on the mean of ECG results corresponding to 3 heart beats.)
* AST<2×upper limit of normal, ALT<2×upper limit of normal, alkaline phosphatase≤1.5×upper limit of normal, bilirubin≤1.5×upper limit of normal at screening (The serum bilirubin shall be fractioned and the direct bilirubin shall be below 35%. In this case, the free bilirubin level exceeding 1.5 times the upper limit of normal is acceptable.)
* Pediatric patients whose parents (persons with parental authority or guardians) shall submit written informed consent
* Pediatric patients whose parents (persons with parental authority or guardians) shall fill the medication diaries

Exclusion Criteria:

* Pediatric patients whose body weight is above or below the infantile growth curves shown in the infant body growth investigation report in 2011 [MHLW, 2011]
* Pediatric patients breast-fed by mothers who take any antihistamine drugs during the study period
* Pediatric patients who received systemic adrenocorticosteroids within 28 days before Visit 2
* Pediatric patients who are currently treated or planned to have immunotherapy initiated during the study period
* Pediatric patients who had abnormal laboratory results that were unrelated to allergic disorders [These patients can be enrolled if the investigator (or sub-investigator) judges that their enrolment poses no clinical problem.]
* Pediatric patients who require application of adrenocorticosteroids for external use that are classified as "strongest," "very strong" or "strong"
* Pediatric patients who suffer from asthma as a complication and require treatment with adrenocorticosteroids (including adrenocorticosteroid combinations)
* Pediatric patients with the history of convulsion, febrile convulsion or sleep apnea
* Pediatric patients whose brothers or sisters have history of sleep apnea or sudden infant death syndrome
* Pediatric patients with history of allergy or hypersensitivity to the ingredients of levocetirizine hydrochloride preparation or piperazine derivatives such as hydroxyzine, cetirizine, cyclizine
* Pediatric patients with history of drug hypersensitivity
* Pediatric patients who are considered inappropriate as the subjects of this clinical trial because of liver diseases, renal diseases, heart diseases or other complications that pose clinical problem
* Pediatric patients whose parents are minors
* Infants who belong to children's institutions
* Pediatric patients who participated in other clinical trials for 6 months before enrolment or those who intend to participate in other clinical trials during the clinical trial period.
* Person meeting any of the following criteria and his/her family (- An employee of GlaxoSmithKline K.K., - Investigator or sub-investigator, - An employee of Site Management Organization (SMO) related with the clinical study)
* Other pediatric patients who are judged as inappropriate for participating in this clinical trial by the investigator (or sub-investigator)

Ages: 6 Months to 23 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2012-04; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- Japan (2):
  - GSK Investigational Site, Chiba
  - GSK Investigational Site, Tokyo

RESULTS

PARTICIPANT FLOW:
Groups:
- Levocetirizine: >=6 Months and <12 Months Old: Participants who were >=6 months and <12 months old received levocetirizine 1.25 milligrams (mg) (2.5 milliliters [mL] as levocetirizine oral solution) once daily in the morning for a duration of 2 weeks.
- Levocetirizine: >=12 Months and <24 Months Old: Participants who were >=12 months and <24 months old received levocetirizine 1.25 mg (2.5 mL as levocetirizine oral solution) twice daily (in the morning and in the evening before going to sleep) for a duration of 2 weeks.
Period: Overall Study
Arm/Group | Levocetirizine: >=6 Months and <12 Months Old | Levocetirizine: >=12 Months and <24 Months Old
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Levocetirizine: >=6 Months and <12 Months Old | Levocetirizine: >=12 Months and <24 Months Old | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: Months] | 8.1 (1.94) | 15.8 (2.56) | 12.0 (4.46)
Gender [Count of Participants; unit: Participants]
  Female | 11 | 17 | 28
  Male | 19 | 13 | 32
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian - Japanese Heritage | 30 | 29 | 59
  Asian - Mixed Race | 0 | 1 | 1
Number of participants with the indicated primary disease at Baseline [Number; unit: participants]
  Allergic rhinitis | 10 | 10 | 20
  Pruritus associated with the skin diseases | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs) and Non-serious Adverse Events (AEs)
Description: A non-serious AE is defined as any untoward medical occurrence in a participant/clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. For marketed medicinal products, this also includes failure to produce expected benefits (i.e., lack of efficacy), abuse, or misuse. An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, or is a possible drug-induced liver injury. For a list of all SAEs/non-serious AEs occurring at a frequency of >=5%, please see the SAE/non-serious AE module of this record.
Time Frame: up to Week 2/Early Withdrawal (EW)
Population: Safety Population : all participants who participated in this study and who received at least one dose of medication
Measure: Number; unit: participants
Groups:
- Levocetirizine: Total Population: Participants received levocetirizine 1.25 mg (2.5 mL as levocetirizine oral solution: once daily for participants who were >=6 months and <12 months old; twice daily for participants who were >=12 months and <24 months old) for a duration of 2 weeks.
Arm/Group | Levocetirizine: >=6 Months and <12 Months Old | Levocetirizine: >=12 Months and <24 Months Old | Levocetirizine: Total Population
Number analyzed (Participants) | 30 | 30 | 60
participants
  Any Adverse Event | 15 | 17 | 32
  Any Serious Adverse Event | 0 | 0 | 0

2. Secondary Outcome: Number of Participants With the Indicated Change From the First Day of Treatment in Allergic Rhinitis and Pruritis Associated With Skin Diseases at Weeks 1 and 2/EW, as Assessed by the Investigator/Sub-investigator Based on Legal Representative Impression
Description: The investigator or sub-investigator made an overall assessment of nasal symptoms (allergic rhinitis [AR]) and pruritus associated with skin diseases (PAWSD) at Weeks 1 and 2 (or at the discontinuation day in the case of early withdrawal [EW] from the clinical trial) by asking the participants' legal representatives to provide feedback using the following scale: 1, significantly improved; 2, moderately improved; 3, mildly improved; 4, no change; 5, mildly worse; 6, moderately worse; 7, significantly worse. Only those participants with AR and PAWSD at Baseline were assessed for improvement in the conditions at Weeks 1 and 2. The "n"s in the category titles reflect the number of participants in the Full Analysis Set (FAS) who had AR and PAWSD at Baseline.
Time Frame: First day of treatment; Weeks 1 and 2/Early Withdrawal
Population: Full Analysis Set (FAS): all participants, excluding those with any major good clinical practice deviation, those who did not meet the primary criteria for enrollment, those who received no dose of study medication, and those with no data after supply of the investigational product
Measure: Number; unit: participants
Arm/Group | Levocetirizine: Total Population
Number analyzed (Participants) | 60
participants
  AR, Week 1, significantly improved, n=20 | 4
  AR, Week 2/EW, significantly improved, n=20 | 8
  AR, Week 1, moderately improved, n=20 | 5
  AR, Week 2/EW, moderately improved, n=20 | 5
  AR, Week 1, mildly improved, n=20 | 4
  AR, Week 2/EW, mildly improved, n=20 | 5
  AR, Week 1, no change, n=20 | 7
  AR, Week 2/EW, no change, n=20 | 1
  AR, Week 1, mildly worse, n=20 | 0
  AR, Week 2/EW, mildly worse, n=20 | 0
  AR, Week 1, moderately worse, n=20 | 0
  AR, Week 2/EW, moderately worse, n=20 | 1
  AR, Week 1, significantly worse, n=20 | 0
  AR, Week 2/EW, significantly worse, n=20 | 0
  PAWSD, Week 1, significantly improved, n=40 | 4
  PAWSD, Week 2/EW, significantly improved, n=40 | 6
  PAWSD, Week 1, moderately improved, n=40 | 11
  PAWSD, Week 2/EW, moderately improved, n=40 | 16
  PAWSD, Week 1, mildly improved, n=40 | 13
  PAWSD, Week 2/EW, mildly improved, n=40 | 14
  PAWSD, Week 1, no change, n=40 | 12
  PAWSD, Week 2/EW, no change, n=40 | 4
  PAWSD, Week 1, mildly worse, n=40 | 0
  PAWSD, Week 2/EW, mildly worse, n=40 | 0
  PAWSD, Week 1, moderately worse, n=40 | 0
  PAWSD, Week 2/EW, moderately worse, n=40 | 0
  PAWSD, Week 1, significantly worse, n=40 | 0
  PAWSD, Week 2/EW, significantly worse, n=40 | 0

3. Secondary Outcome: Number of Participants With the Indicated Change From the First Day of Treatment in Nasal Symptoms and Pruritis Associated With Skin Diseases at Weeks 1 and 2/Early Withdrawal, as Assessed by the Investigator or Sub-investigator
Description: The investigator or sub-investigator comprehensively assessed the participants' improvement in nasal symptoms (allergic rhinitis [AR]) and pruritus associated with skin diseases (PAWSD) at Weeks 1 and 2 (or at the discontinuation day in the case of early withdrawal [EW] from the clinical trial) compared to the first day of treatment by using the following scale: 1, markedly improved; 2, moderately improved; 3, slightly improved; 4, no change; 5, worsened.
Time Frame: First day of treatment; Weeks 1 and 2/Early Withdrawal
Population: FAS. Only those participants with AR and PAWSD at Baseline were assessed for improvement in the conditions at Weeks 1 and 2/Early Withdrawal. The "n"s in the category titles reflect the number of participants in the Full Analysis Set (FAS) who had AR and PAWSD at Baseline.
Measure: Number; unit: participants
Groups:
- Levocetrizine: Total Population: Participants received levocetirizine 1.25 mg (2.5 mL as levocetirizine oral solution: once daily for participants who were >=6 months and <12 months old; twice daily for participants who were >=12 months and <24 months old) for a duration of 2 weeks.
Arm/Group | Levocetrizine: Total Population
Number analyzed (Participants) | 60
participants
  AR, Week 1, markedly improved, n=20 | 7
  AR, Week 2/EW, markedly improved, n=20 | 12
  AR, Week moderately improved, n=20 | 4
  AR, Week 2/EW, moderately improved, n=20 | 3
  AR, Week 1, slightly improved, n=20 | 3
  AR, Week 2/EW, slightly improved, n=20 | 4
  AR, Week 1, no change, n=20 | 6
  AR, Week 2/EW, no change, n=20 | 1
  AR, Week 1, worsened, n=20 | 0
  AR, Week 2/EW, worsened, n=20 | 0
  PAWSD, Week 1, markedly improved, n=40 | 6
  PAWSD, Week 2/EW, markedly improved, n=40 | 10
  PAWSD, Week 1, moderately improved, n=40 | 15
  PAWSD, Week 2/EW, moderately improved, n=40 | 19
  PAWSD, Week 1, slightly improved, n=40 | 12
  PAWSD, Week 2/EW, slightly improved, n=40 | 8
  PAWSD, Week 1, no change, n=40 | 7
  PAWSD, Week 2/EW, no change, n=40 | 3
  PAWSD, Week 1, worsened, n=40 | 0
  PAWSD, Week 2/EW, worsened, n=40 | 0

4. Secondary Outcome: Number of Participants Categorized With the Indicated Pruritis Severity on the First Day of Treatment and at Weeks 1 and 2/Early Withdrawal
Description: The investigator comprehensively assessed the pariticipant's severity of pruritus on the first day of treatment (FDOT), at Week 1, and at Week 2 (or at the discontinuation day in the case of early withdrawal [EW] from the clinical trial) by using the following scale: 4, severe; 3, moderate; 2, mild; 1, slight; 0, none.
Time Frame: First day of treatment; Weeks 1 and 2/Early Withdrawal
Population: FAS. Only those participants with pruritis associated with skin diseases at Baseline were assessed for pruritis severity.
Measure: Number; unit: participants
Arm/Group | Levocetrizine: Total Population
Number analyzed (Participants) | 40
participants
  FDOT, none | 0
  FDOT, slight | 7
  FDOT, mild | 17
  FDOT, moderate | 11
  FDOT, severe | 5
  Week 1, none | 6
  Week 1, slight | 14
  Week 1, mild | 11
  Week 1, moderate | 7
  Week 1, severe | 2
  Week 2/EW, none | 13
  Week 2/EW, slight | 8
  Week 2/EW, mild | 11
  Week 2/EW, moderate | 8
  Week 2/EW, severe | 0

5. Secondary Outcome: Cmax and Cmin of Levocetirizine in Plasma
Description: Cmax is defined as the peak plasma concentration of a drug after administration. Cmin is defined as the lowest (trough) concentration that a drug reaches before the next dose is administered. For both age cohorts, blood samples were collected 1.5-2.5 hours after the last drug administration for assessment of Cmax at either Week 1 or 2/EW. For participants in the >=6 months and <12 months cohort, blood samples were collected 22.5-25.5 hours after the last drug administration for Cmin at a different visit from Cmax sampling. For participants in the >=12 months and <24 months cohort, blood samples were collected 10.5-13.5 hours after the final drug administration for Cmin at a different visit from Cmax sampling. For all participants, if Cmin sampling occurred at Week 1, then Cmax sampling occurred at Week 2/EW, and vice versa.
Time Frame: Weeks 1 and 2/Early Withdrawal
Population: Pharmacokinetic Concentration Population: all participants who underwent blood sampling, who provided data at the time of the last dose and the time of blood sampling, and who provided valid drug concentrations
Measure: Median (Full Range); unit: nanograms per milliliter
Arm/Group | Levocetirizine: >=6 Months and <12 Months Old | Levocetirizine: >=12 Months and <24 Months Old
Number analyzed (Participants) | 30 | 30
nanograms per milliliter
  Cmax | 206.780 [41.89 to 327.03] | 213.440 [17.75 to 323.42]
  Cmin | 17.710 [3.49 to 104.46] | 48.330 [2.91 to 126.18]

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious AEs were collected from the start of the study up to Week 2/Early Withdrawal.
Description: SAEs and non-serious AEs were collected in members of the Safety Population, comprised of all participants who received at least one dose of study medication.
Arm/Group | Levocetirizine: >=6 Months and <12 Months Old | Levocetirizine: >=12 Months and <24 Months Old | Levocetirizine: Total Population
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/60
Other Adverse Events (participants affected / at risk) | 7/30 | 12/30 | 19/60
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Levocetirizine: >=6 Months and <12 Months Old (N=30) | Levocetirizine: >=12 Months and <24 Months Old (N=30) | Levocetirizine: Total Population (N=60)
Nasopharyngitis (Infections and infestations) | 0 | 7 | 7
Gastroenteritis (Infections and infestations) | 1 | 2 | 3
Diarrhoea (Gastrointestinal disorders) | 2 | 2 | 4
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 3
Eczema (Skin and subcutaneous tissue disorders) | 2 | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.